CLINICAL TRIAL: NCT03244683
Title: A Study of the Efficacy of Oral Nutritional Supplementation to Reduce Postoperative Complications Associated With Pancreatic Surgery
Brief Title: A Study of the Efficacy of ONS to Reduce Postoperative Complications Associated With Pancreatic Surgery
Acronym: INSPIRE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to low enrollment
Sponsor: Ohio State University (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Principal Investigator, Philip Hart, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0170
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Subjects randomized to this arm will receive: An Oral Nutritional Supplementation (Ensure Surgical), home-based resistance training, and dietary counseling
  Interventions: Dietary Supplement: Ensure Surgical; Other: Nutrition counseling; Other: Low-intensity exercise therapy
- Nutrition Counseling alone (Other): Subjects randomized to this arm will receive: Dietary counseling along with standard of care procedures.
  Interventions: Other: Nutrition counseling

INTERVENTIONS:
Dietary Supplement: Ensure Surgical — Subjects randomized to the intervention arm will consume two Ensure Surgical for 5-7 days.
  Arms: Intervention
Other: Nutrition counseling — All study subjects will be provided with nutrition counseling at the time of study enrollment.
Other: Low-intensity exercise therapy — Patients randomized to the intervention arm will also be provided with verbal and written instructions for light resistance training. The exercises will be performed at home during the preoperative study period.
  Arms: Intervention

SUMMARY:
This is a single center, open label, randomized trial, involving 150 patients undergoing pancreatic surgery. Patients will be randomized at the time of enrollment to receive from 5-7 days of ONS supplementation combined with resistance training and nutritional education compared to standard of care, consisting of nutritional education alone.

This proof of concept study is intended to demonstrate the ability of pre-habilitation to improve patient-related outcomes following pancreatic surgery, specifically postoperative complications. The rationale for using the designated oral nutrient supplementation is to preserve muscle mass, and decrease weight loss.

DETAILED DESCRIPTION:
Patients undergoing pancreatic surgery for either chronic pancreatitis or known/suspected pancreatic cancer represent the study population for this clinical trial.

Study subjects randomized to one of the ONS arms will be asked to consume the drink during the study intervention. Study visits immediately preoperative, and 1, 3, and 6 months following surgery will be in-person visits. If subjects are unable to return to our Institution for subsequent clinical care, these telephone interviews will be collected and acquisition of locally obtained laboratory tests will be attempted.

Assessments performed during postoperative visits include:

* Vital signs and physical examination
* Blood samples
* Performance status and strength
* Quality of life measures
* Postoperative complications and hospital readmissions (if any)

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-89 at the time of study enrollment.
2. Undergoing pancreatectomy for either chronic pancreatitis or pancreatic cancer.
3. Ability and willingness to complete study related documents and activities.

Exclusion Criteria:

1. Severe malnutrition that in the judgment of the patient's supervising physician or an investigator would not permit surgical intervention without preoperative nutritional support (enteral or parenteral).
2. Subject is receiving (or planned to receive) enteral tube feeding or parenteral nutrition at the time of screening or before surgery.
3. Surgery is planned within 7 days of enrollment (i.e., inadequate time to offer the study intervention).
4. Known allergy to soy or milk, which are included in the oral supplement.
5. The inability to refrain from using a non-study oral nutritional supplement or fish oil supplementation (unless prescribed for treatment of hyperlipidemia).
6. Pregnancy, incarceration, or inability to provide written informed consent.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  The postoperative complication rate of 1 or more complication

SECONDARY OUTCOMES:
Supplement compliance | 7-14 days
  Frequency of subjects compliant with ≥70% of the provided preoperative supplement.
Anthropometric measures | 30 days
  Serial anthropometric measures.
Length of stay and readmission | 30 days
  Hospital length of stay and readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Philip Hart, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers.